CLINICAL TRIAL: NCT02694809
Title: A Large-scale Multicenter Phase II Study Evaluating the Protective Effect of a Tissue Selective Estrogen Complex (TSEC) in Women With Newly Diagnosed Ductal Carcinoma in Situ
Brief Title: The PROMISE Study: Duavee in Women With DCIS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Pfizer (Industry); University of Chicago - Department for Cancer Research (Unknown); University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NU 15B06; STU00202100 (CTRP (Clinical Trial Reporting Program)); NU 15B06 (Other: Northwestern University); P30CA060553 (NIH); NCI-2016-00066 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2016-02-24; First posted 2016-03-01 (Estimated); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Ductal Breast Carcinoma In Situ; Postmenopausal
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating | interventions — Estrogens, Conjugated (USP); bazedoxifene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (conjugated estrogens/bazedoxifene) (Experimental): Patients receive conjugated estrogens/bazedoxifene orally (PO) once daily (QD) for 28 +/- 7 days in the absence of disease progression or unacceptable toxicity. Patients then undergo surgery.
  Interventions: Drug: Conjugated Estrogens/Bazedoxifene; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Procedure: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (placebo) (Placebo Comparator): Patients receive placebo PO QD for 28 +/- 7 days in the absence of disease progression or unacceptable toxicity. Patients then undergo surgery.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Other: Placebo; Procedure: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Conjugated Estrogens/Bazedoxifene — Given PO
  Arms: Arm I (conjugated estrogens/bazedoxifene)
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Other: Placebo — Given PO
  Other Names: placebo therapy; PLCB; sham therapy
  Arms: Arm II (placebo)
Procedure: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
The main purpose of this study is to determine if taking the study drug, conjugated estrogens/bazedoxifene (Duavee®) causes any changes in the proliferation markers within the breast tissue of the study subjects. The study drug is approved by the US Food and Drug Administration in healthy postmenopausal women to treat certain symptoms of menopause such as hot flashes. Since it is not approved in women with DCIS, its use in this study is experimental. This study will also look at whether taking the study drug causes any significant or undesirable side effects in women with DCIS. The researchers hope that this study will help them determine if taking the study drug is safe in women taking DCIS and if it can possibly reduce the risk of developing breast cancer in women with DCIS.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES;

• To determine if CE/BZA reduces proliferation as measured by Ki-67 protein expression

Secondary Objectives:

* To determine if CE/BZA modulates expression of ERα, progesterone receptor (PR) and human epidermal growth factor receptor 2 (HER-2).
* To determine if CE/BZA modulates a previously validated set of epithelial markers of progression.
* To determine if TSECs will restore expression of the stromal marker CD36 and repress pro-tumorigenic ECM proteins and soluble factors.
* To determine if a short intervention with CE/BZA results in any difference in Quality of Life (QOL) as it relates to menopausal symptoms in postmenopausal women with DCIS.
* To determine if a short intervention with CE/BZA has a favorable side effect profile compared with other endocrine therapy interventions using the validated Breast Cancer Prevention Trial Eight Symptom Scale (BESS) questionnaire.

Exploratory Objectives

* To determine if CE/BZA alters expression of estrogen-modulated genes and elicits novel ER dependent-gene signatures in breast epithelium
* To demonstrate that CE/BZA does not upregulate Anterior Gradient 2 (AGR2), a marker of ERα agonist activity.
* To determine if CE/BZA will modulate some aspects of immune function as measured by a switch to a M2-type pro-tumorigenic macrophage signature and an immunosuppressive T cell signature.
* To determine if a short intervention with CE/BZA alters expression of estrogen-modulated genes and elicits novel ER dependent-gene signatures in the breast stroma.
* To determine if CE/BZA affects plasma concentrations of BZA in patients with the UGT1A1*28 gene polymorphism.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive conjugated estrogens/bazedoxifene orally (PO) once daily (QD) for 28 +/- 7 days in the absence of disease progression or unacceptable toxicity. Patients then undergo surgery.

ARM II: Patients receive placebo PO QD for 28 +/- 7 days in the absence of disease progression or unacceptable toxicity. Patients then undergo surgery.

ELIGIBILITY:
Inclusion Criteria:

* Women must have newly diagnosed histologically confirmed ER (+) DCIS scheduled to undergo surgical therapy. The pathology report (signed pathology report from attending pathologist) from each individual institution will be used to determine eligibility. Extent of DCIS in imaging per site institutional standard.

Note: After the patient has completed the study and the slides have been sent to NU, our pathologists will review the slides to confirm the diagnosis.

Note: DCIS suspicious for micro invasion is eligible on core biopsy. This is due to the fact that many these patients will not have invasion on final pathology.

Note: Women presenting with bilaterial DCIS are eligible but if both right and left DCIS are ER+, we will only accept tissue from the side with the largest area of DCIS based on imaging and pathology criteria outlined later in the protocol.

* DCIS must be ≥ 1cm based on extent of calcifications, presence of a mass on ultrasound OR enhancement on MRI OR DCIS must be ≥ 5mm of DCIS on one single core. Can be < 5mm if DCIS is identified on multiple cores (at least 2 cores)
* Women presenting after excision with positive margins are eligible. Ki-67, Cox-2, P-16, expression in immediately adjacent tissue is similar to what is found in DCIS.

Note: Positive margins are defined as DCIS present at the inked margin or DCIS <1mm from the margin. - Women must be postmenopausal (defined as no menstrual cycle for 12 months or surgical history of bilateral salpingoopherectomy. Postmenopausal women of all races and ethnic groups are eligible to participate for this trial. Men are not eligible.

Note: women who have had a hysterectomy without a bilateral salpingoopherectomy may still be pre-menopausal. Confirmation of postmenopausal status is required for these patients and will be measured by testing levels of estradiol, progesterone and FSH (lab ranges per institutional standards). In addition, confirmation of postmenopausal status may be performed in any patient with unclear menopausal status per treating physician discretion.

* Women in the age range of ≥18-79 (inclusive)
* ECOG performance status ≤ 2 (Karnofsky ≥60%, see Appendix A).
* Patients must have normal organ and marrow function as defined below Leukocytes ≥3,000/mcL Platelets ≥100,000/mcL Hemoglobin ≥ 9g/dl Total Bilirubin ≤ 1.5 x upper limit of normal (ULN) AST (SGOT) and ALT (SGPT)

  * 2.5 × institutional upper limit of normal Serum Creatinine OR Creatinine Clearance
  * 1.5 x ULN ≥60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal (calculated with the Cockcroft-Gault Equation in EPIC)
* Patients must have the ability to swallow oral medication
* Ability to understand and the willingness to sign a written informed consent document and comply with all procedures

Exclusion Criteria

* Patients who are receiving any other investigational agents. A minimum of 4 weeks wash-out period is required for eligibility. Please contact Principal Investigator, Dr. Swati Kulkarni for further clarification
* Patients with a "currently active" second malignancy other than non-melanoma skin cancers. Patients are not considered to have a "currently active" malignancy if they have completed therapy and are free of disease for ≥ 1 years.
* History of allergic reactions/hypersensitivity attributed to compounds of similar chemical or biologic composition to CE/BZA. (I.e. same class of drug as CE/BZA)
* Current HRT, SERM or Aromatase Inhibitor (AI) use. If yes, the wash-out period is 30 days before diagnostic core needle biopsy.

Note: Local therapy (i.e. estrogen cream) will be permitted due to low systemic absorption of estrogen. Note: if patient is registered prior to completed washout, diagnostic core needle biopsy date will need to be provided.

* Confirmed current of invasive breast cancer Note: Patients who do not currently have a diagnosis of invasive breast cancer but who are planning to undergo additional standard of care testing to rule out a diagnosis of invasive breast cancer (such as future imaging or biopsy) are eligible. If the results of this standard of care testing later confirm that the subject has a diagnosis of invasive breast cancer, the subject should be withdrawn from the study at that time.
* Patients with recurrent ipsilateral DCIS
* Any of the following conditions, or a known history of any of the following:

  * deep venous thrombosis,
  * pulmonary embolism,
  * retinal vascular thrombosis,
  * any arterial thrombosis,- Known protein C, protein S, or anti-thrombin deficiency or other known thrombophilic disorders including stroke and myocardial infarction
* Unexplained/undiagnosed abnormal uterine bleeding (concern for undiagnosed endometrial cancer)
* Women who are pregnant or lactating. CE/BZA may cause fetal harm when administered to a pregnant woman. If this drug is used during pregnancy, or if the patient becomes pregnant while taking this drug, the patient should be apprised of the potential hazard to a fetus.
* Patients receiving any medications or substances that are strong inhibitors or inducers of CYP3A4 and UGT are ineligible. The wash out period for such drugs is a minimum of 7 days or 5 half-lives whichever is shorter. Refer to Appendix C.

Note: As this list is constantly evolving, if a medication is incorrectly documented as prohibited in this protocol, documentation from the site pharmacist to the contrary will be acceptable for the purposes of registration.

- Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Ages: 18 Years to 79 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2017-01; Primary Completion 2024-06-19 (Actual); Study Completion 2024-06-19 (Actual)

PRIMARY OUTCOMES:
Change in Ki-67 protein expression | Up to 5 weeks
  Evaluating if CE/BZA reduces proliferation as measured by Ki-67 protein expression. Change in Ki-67 between baseline and end of the intervention will be measured.

SECONDARY OUTCOMES:
Expression of ERα | Up to 5 weeks
  Determine if CE/BZA modulates expression of ERα.
Expression of progesterone receptor (PR) | Up to 5 weeks
  Evaluate if CE/BZA modulates expression of PR
Expression of human epidermal growth factor receptor 2 (HER-2) | Up to 5 weeks
  Determine if CE/BZA modulates expression of HER-2.
Epithelial markers of progression | Up to 5 weeks
  Evaluate if CE/BZA modulates a previously validated set of epithelial markers of progression.
Expression of the stromal marker CD36 | Up to 5 weeks
  Determine if TSECs will restore expression of the stromal marker CD36.
Repression of pro-tumorigenic ECM proteins | Up to 5 weeks
  Determine if TSECs will repress pro-tumorigenic ECM proteins.
Repression of soluble factors | Up to 5 weeks
  Determine if TSECs will repress soluble factors.
Quality of Life (QOL) | Up to 5 weeks
  Evaluate if a short intervention with CE/BZA results in any difference in Quality of Life (QOL) as it relates to menopausal symptoms in postmenopausal women with DCIS.
Breast Cancer Prevention Trial Eight Symptom Scale (BESS) questionnaire | Up to 5 weeks
  Determine if a short intervention with CE/BZA has a favorable side effect profile compared with other endocrine therapy interventions using the validated Breast Cancer Prevention Trial Eight Symptom Scale (BESS) questionnaire.

OTHER OUTCOMES:
Expression of estrogen-modulated genes in breast epithelium | Up to 5 weeks
  Determine if CE/BZA alters expression of estrogen-modulated genes in breast epithelium.
Novel ER dependent-gene signatures in breast epithelium | Up to 5 weeks
  Evaluate if CE/BZA elicits novel ER dependent-gene signatures in breast epithelium.
Anterior Gradient 2 (AGR2) | Up to 5 weeks
  Demonstrate that CE/BZA does not upregulate Anterior Gradient 2 (AGR2), a marker of ERα agonist activity.
M2-type pro-tumorigenic macrophage signature | Up to 5 weeks
  Determine if CE/BZA will modulate some aspects of immune function as measured by a switch to a M2-type pro-tumorigenic macrophage signature.
Immunosuppressive T cell signature | Up to 5 weeks
  Determine if CE/BZA will modulate some aspects of immune function as measured by a switch to a an immunosuppressive T cell signature.
Estrogen-modulated genes in the breast stroma | Up to 5 weeks
  Evaluate if a short intervention with CE/BZA alters expression of estrogen-modulated genes in the breast stroma.
Novel ER dependent-gene signatures in the breast stroma | Up to 5 weeks
  Determine if a short intervention with CE/BZA elicits novel ER dependent-gene signatures in the breast stroma.
plasma concentrations of BZA | Up to 5 weeks
  Evaluate if CE/BZA affects plasma concentrations of BZA in patients with the UGT1A1*28 gene polymorphism.

CONTACTS AND LOCATIONS:
Overall Officials: Swati Kulkarni, MD, Principal Investigator — Northwestern University
Locations (10):
- United States (10):
  - University of Colorado at Denver/ Department of Surgery, Aurora, Colorado
  - Northwestern University, Chicago, Illinois
  - Northwestern Medicine - Delnor/Warrenville Cancer Centers/Central DuPage Hospital, Geneva, Illinois
  - Northwestern University, Lake Forest, Illinois
  - John's Hopkins University, Baltimore, Maryland
  - Dana Farber/Partners Cancer Care Inc, Boston, Massachusetts
  - Washington University in St. Louis/ Siteman Cancer Center, St Louis, Missouri
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Pittsburg/ Magee-Womens Hospital, Pittsburgh, Pennsylvania
  - Huntsman Cancer Institute, Salt Lake City, Utah